CLINICAL TRIAL: NCT05059847
Title: Impact of Cross-training on Induction Treatment Response in Acute Lymphoblastic Leukemia Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Christian Omar Ramos-Peñafiel, MD, PhD, Principal Investigator, Hospital General de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HGMDI/21/204/03/46
Record Dates: First submitted 2021-09-07; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Acute Lymphoblastic Leukemia, Adult B-Cell
Keywords: Acute lymphoblastic leukemia; Interleukine-15; Cross-training; Body Composition; Physical performance
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Clinical randomized single blinded trial
Who Masked: Investigator
Masking Description: The masking of the study will be for the principal investigator, only knowing the maneuver person in charge of the routine and the patient. The patients who will practice the exercise intervention will be carry out in certain space and time that does not interfere with the medical intervention and in which the treating medical personnel will not be present.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care Group (No Intervention): Each patient will receive the standard pharmacological treatment for patients with Acute Lymphoblastic Leukemia based on 3 cycles of chemotherapy (21 days duration per cycle); plus the World Health Organization recommendation that indicates at least 150 min a week of moderate physical activity, equivalent to walking 30 minutes a day for 5 days at an intensity between 60 and 70% of your maximum heart rate.
- Resistance Training Group (Active Comparator): Each patient will receive the standard pharmacological treatment for patients with Acute Lymphoblastic Leukemia based on 3 cycles of chemotherapy (21 days duration per cycle); plus a resistance exercise routine using weights. An individualized program with exercises supervised by a trainer and basic medical team will be developed for each patient during their hospital stay. Each training routine will have a monthly exercise progression based on intensity, frequency and / or duration.
  Interventions: Other: Training
- Cross-training Group (Experimental): Each patient will receive the standard pharmacological treatment for patients with Acute Lymphoblastic Leukemia based on 3 cycles of chemotherapy (21 days duration per cycle); plus a cross-training routine using implements without any extra weight to improve stability, joint mobility and general strength of the body. An individualized program with exercises supervised by a trainer and basic medical team will be developed for each patient during their hospital stay. Each training routine will have a monthly exercise progression based on intensity, frequency and / or duration.
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — Training routine assigned by randomized chart
  Arms: Cross-training Group; Resistance Training Group

SUMMARY:
Despite advances in the treatment of acute lymphoblastic leukemia, the prognosis in adults is still poor, largely due to the resistance of treatment at diagnosis or early relapse. Among the strategies associated with the treatment of Acute Lymphoblastic Leukemia is rehabilitation and physical medicine in order to improve the quality of life, body composition, fitness, strength and improve the attachment and acceptance of their treatment

DETAILED DESCRIPTION:
Previous evidence had shown that among the beneficial effects of an exercise intervention in cancer is the reduction of adverse events associated with treatment, such as nausea and fatigue. Also, the overexpression of Interleukin-15 in cancer is related to a poor prognosis, biologically the implementation of a cross-training exercise routine can function as a regulatory pathway for its expression due to its consumption at muscular level. Finally, the time to consider a relapse with a very poor prognosis is during first three months of treatment, so implementation of an exercise strategy during this period could reduce the proportion of early relapses mediated by Interleukin-15 expression

ELIGIBILITY:
Inclusion Criteria:

* Ability to walk without support.
* Life expectancy greater than 7 days
* Previous authorization of treating hematologist for participation
* Acceptance and signing of informed consent form

Exclusion Criteria:

* Patients with neutropenia, infections and / or bleeding on admission to hospitalization.
* Patients that are unable to perform physical activity.
* Central nervous system diseases that make movement impossible.
* Cardiac function alterations assessed by electrocardiogram and echocardiogram
* Patients in relapse
* Patients referred from another hospital and who are been attended in our hospital

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-01-13 (Estimated); Study Completion 2023-05-19 (Estimated)

PRIMARY OUTCOMES:
Interleukin 15 | 3 months
  Pro-inflammatory cytokine concentration, measured through peripheral blood
Neutrophils count | 3 months
  Number of neutrophils found in peripheral blood at the end of each chemotherapy cycle
Luekocytes count | 3 months
  Number of leukocytes found in peripheral blood at the end of each chemotherapy cycle
Platelets count | 3 months
  Number of platelets found in peripheral blood at the end of each chemotherapy cycle
Hemoglobin count | 3 months
  Number of hemoglobin found in peripheral blood at the end of each chemotherapy cycle
Functional Assessment of Cancer Therapy- Leukemia | 3 months
  Psychological test that evaluates quality of life from four different areas: functional, emotional, social and physical wellness.
Blasts in marrow | 3 months
  Presence of more than 20% of blasts in bone marrow after each chemotherapy cycle.

SECONDARY OUTCOMES:
Complications during hospital stay | 1 month
  Presence or absence of complications during the hospital stay, for example: neutropenic fever, infections, severe mucositis and/or cardiotoxicity.
Admission to ICU | 3 months
  Admission to ICU during the protocol
Hospital Stay | 1 month
  Measurement of days of hospital stay
Hospital Discharge | 3 months
  The event in which patient is dishcarge from Hopital stay,

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Martinez Tovar, PhD, Study Director — Hospital General de Mexico
Locations (1):
- Hospital General de México "Dr. Eduardo Liceaga", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
All participants and its information will be managed by intern investigators and will be kept secure for personal data protection according to Mexican laws

REFERENCES:
- [Background] Gomez-Almaguer D, Marcos-Ramirez ER, Montano-Figueroa EH, Ruiz-Arguelles GJ, Best-Aguilera CR, Lopez-Sanchez MD, Barrera-Chairez E, Lopez-Arrollo JL, Ramos-Penafiel CO, Leon-Pena A, Gonzalez-Lopez EE, Rivas-Garcia PE, Tellez-Hinojosa CA, Gomez-De Leon A, Jaime-Perez JC. Acute Leukemia Characteristics are Different Around the World: the Mexican Perspective. Clin Lymphoma Myeloma Leuk. 2017 Jan;17(1):46-51. doi: 10.1016/j.clml.2016.09.003. Epub 2016 Sep 17. PMID 27742477
- [Background] Alibhai SM, Durbano S, Breunis H, Brandwein JM, Timilshina N, Tomlinson GA, Oh PI, Culos-Reed SN. A phase II exercise randomized controlled trial for patients with acute myeloid leukemia undergoing induction chemotherapy. Leuk Res. 2015 Aug 28:S0145-2126(15)30365-9. doi: 10.1016/j.leukres.2015.08.012. Online ahead of print. PMID 26350143
- [Result] Coombs A, Schilperoort H, Sargent B. The effect of exercise and motor interventions on physical activity and motor outcomes during and after medical intervention for children and adolescents with acute lymphoblastic leukemia: A systematic review. Crit Rev Oncol Hematol. 2020 Aug;152:103004. doi: 10.1016/j.critrevonc.2020.103004. Epub 2020 May 27. PMID 32580035